CLINICAL TRIAL: NCT06212401
Title: Comparison of Dexmedetomidine Versus Ketofol For Moderate Sedation In Endoscopic Retrograde Cholangiopancreatography (ERCP): A Randomized Controlled Trial
Brief Title: Dexmedetomidine Versus Ketofol for Moderate Sedation in Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Syed Muhammad Abbas, Principal Investigator, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 234
Record Dates: First submitted 2023-12-23; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine in a 2 ml ampule of 100 ug/ml diluted in 18 ml of normal saline, making a total volume of 20 ml.
  Interventions: Drug: Dexmedetomidine
- Ketofol (Active Comparator): 2 ml ketamine (50mg/ml) and 10 ml of propofol 1% (10mg/ml) diluted in 8 ml of normal saline. This mixture was 20 ml each, making 5mg/ml of ketamine and propofol.
  Interventions: Drug: Ketofole

INTERVENTIONS:
Drug: Dexmedetomidine — Patients received dexmedetomidine as a bolus over 10 minutes in a dose of 1ug/kg followed by an infusion at the rate of 0.5ug/kg/hr
  Arms: Dexmedetomidine
Drug: Ketofole — Patients received ketofol 1mg/kg over 10 minutes followed by 50ug/kg/min of infusion
  Arms: Ketofol

SUMMARY:
Patients were randomly divided into Dexmedetomidine or Ketofol for sedation. In patients who received Dexmedetomidine, a 2ml ampule of 100 ug/ml was diluted in 18 ml of normal saline, making a total volume of 20 ml. Patients received dexmedetomidine as a bolus over 10 minutes in a dose of 1ug/kg followed by an infusion at the rate of 0.5ug/kg/hr and it was labeled as "infusion 1". In the Ketofol group, 2 ml ketamine (50mg/ml) and 10 ml of propofol 1% (10mg/ml) were diluted in 8ml of normal saline. This mixture was 20 ml each, making 5mg/ml of ketamine and propofol. Patients received 1mg/kg over 10 minutes followed by 50ug/kg/min of infusion, labeled as "infusion 2".

DETAILED DESCRIPTION:
Patients aged 20-60 years of any gender scheduled for elective ERCP were included. All these patients had American Society of Anesthesiologists (ASA) classification I or II. While those who were allergic to dexmedetomidine, Ketofol, or related medications, BMI over 36 kg/m2 (morbidly obese), had a history of stroke, renal impairment, chronic obstructive pulmonary disease, asthma, chronic liver disease, hypothyroidism, and congestive cardiac failure were excluded. Furthermore, pregnant, or breastfeeding women or patients who reported chronic use of sedative medications or substance abuse, known contraindications to ERCP, and already enrolled in another clinical trial study were excluded.

Patients were randomly divided into two groups using computer randomization. All patients were taken to the procedure room and venous access was secured on a non-dominant hand by 20G IV cannula, intravenous (I/V) fluid (ringer lactate or normal saline) was started by 8 ml/kg/h, and oxygen support was provided by nasal cannula at 4 liters per minute. Standard monitors were attached for heart rate (HR), noninvasive blood pressure (systolic and diastolic), mean arterial blood pressure (MAP), and peripheral oxygen saturation SpO2. Injection midazolam 0.05 mg/kg was also given I/V to every patient in both groups to decrease the anxiety of patients.

Patients received either Dexmedetomidine or Ketofol for sedation. All syringes and infusion sets were covered by silver paper and these infusions were labeled as infusion 1 or 2. In patients who received Dexmedetomidine, a 2ml ampule of 100 ug/ml was diluted in 18 ml of normal saline, making a total volume of 20 ml. Patients received dexmedetomidine as a bolus over 10 minutes in a dose of 1ug/kg followed by an infusion at the rate of 0.5ug/kg/hr and it was labeled as "infusion 1". In the Ketofol group, 2 ml ketamine (50mg/ml) and 10 ml of propofol 1% (10mg/ml) were diluted in 8ml of normal saline. This mixture was 20 ml each, making 5mg/ml of ketamine and propofol. Patients received 1mg/kg over 10 minutes followed by 50ug/kg/min of infusion, labeled as "infusion 2".

During infusion, vitals were recorded at 0,1,3,5, and 10-minute intervals from the start, and the Ramsay Sedation scale score (RSS) was recorded every 1 minute. Both infusions were started as per the randomization of groups. The mean difference in time to achieve adequate sedation and time to good recovery were noted as outcomes in each group. In addition, complications during the procedure and recovery were also noted. Adequate sedation was defined as the time from initiation of infusion to achieve an RSS score of 4. While Modified Aldrete's score (MAS) was used to assess the recovery. Time from discontinuation of the infusion to achieve an MAS score of 9 was labeled as a good recovery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-60 years
* Any gender
* Scheduled for elective ERCP
* American Society of Anesthesiologists (ASA) classification I or II

Exclusion Criteria:

* Allergic to dexmedetomidine, Ketofol, or related medications
* BMI over 36 kg/m2 (morbidly obese)
* History of stroke, renal impairment, chronic obstructive pulmonary disease, asthma, chronic liver disease, hypothyroidism, and congestive cardiac failure

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Ramsay sedation score | 0-2 hours
  Clinical Score Patient's Characteristics
  1. Awake; agitated or restless or both
  2. Awake; cooperative, oriented, and tranquil
  3. Awake but responds to commands only
  4. Asleep; brisk response to light glabellar tap or loud auditory stimulus
  5. Asleep; sluggish response to light glabellar tap or loud auditory stimulus
  6. Asleep; no response to glabellar tap or loud auditory stimulus

SECONDARY OUTCOMES:
Modified Aldrete's score | 10-15 minutes
  Modified Aldrete's Score, also known as the Aldrete Score, consists of five criteria, each scored from 0 to 2, with a maximum total score of 10. The criteria are:
  1. Activity
  2. Respiration
  3. Circulation
  4. Consciousness
  5. Oxygen Saturation
     * A score of 9-10 indicates the patient is ready for discharge from the recovery area.
     * A score of 8 may be acceptable for discharge based on the surgeon's and anesthetist's discretion.
     * Scores below 8 may necessitate further observation and interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Syed M Abbas, FCPS, Principal Investigator — Sindh Institute of Urology and Transplantation
Locations (1):
- Sindh Institute of Urology and Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT06212401/Prot_SAP_ICF_000.pdf